CLINICAL TRIAL: NCT00098137
Title: Angiotensin II-Antagonist in Paroxysmal Atrial Fibrillation Trial (ANTIPAF Trial)
Brief Title: Trial to Investigate the Efficacy of Olmesartan in Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFNET-B10; Grant No 01GI0204 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Heart Disease; Arrhythmia; Atrial Fibrillation
Keywords: atrial fibrillation; angiotensin II; angiotensin receptor antagonist; drug; controlled clinical trial
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Atrial Fibrillation | interventions — olmesartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olmesartan (Experimental): Olmesartan tablet, 1 in the morning
  Interventions: Drug: Olmesartan
- Placebo (Placebo Comparator): Placebo tablets, 1 in the morning
  Interventions: Drug: Olmesartan

INTERVENTIONS:
Drug: Olmesartan

SUMMARY:
Hypothesis:

Blocking the angiotensin (AT) II type 1 receptor (Olmesartan) reduces the incidence of episodes of atrial fibrillation in patients with paroxysmal atrial fibrillation during 12 months by more than 25% compared to standard medication without angiotensin II type 1 receptor.

A total of 422 subjects will be included in the two study groups. The treatment arm will receive 40mg Olmesartan per day, the remaining patients will receive placebo. Follow-up is 12 months. Daily Tele-ECG recordings will determine the cardiac rhythm and asymptomatic episodes of atrial fibrillation (AF) every day. Concomitant therapy with AV-nodal blocking drugs are allowed during the study. In case of severe AF-induced symptoms, an antiarrhythmic "recovery medication" (amiodarone) is allowed during follow-up.

DETAILED DESCRIPTION:
Double-blind, central randomization, two treatment groups, stratified by beta-blocker use. 211 patients in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal atrial fibrillation: ECG documentation of atrial fibrillation at least in one ECG recorded during the last 2 months prior to randomization plus additional ECG recording of sinus rhythm at least 12 hours after the above mentioned ECG documentation.
* Age ≥ 18
* Patient informed orally and in writing
* Written informed consent of the patient

Exclusion Criteria:

* Strong clinical evidence for therapy with AT II/ACE inhibitors
* AT II/ACE inhibitor therapy within the last month
* Therapy with antiarrhythmic agents of class I or class III within the last month, therapy with amiodarone within the last 3 months
* Direct current (DC) cardioversion within the last 3 months
* Symptomatic bradycardia
* Implanted pacemaker or implanted cardioverter/defibrillator with any antitachycardiac algorithm in use
* Cardiac surgery or cardiac catheter ablation within the last 3 months
* Typical angina pectoris symptoms at rest or during exercise
* Known coronary artery disease with indication for intervention
* Valvular disease > II degree
* Left ventricular ejection fraction < 40%
* Diastolic blood pressure > 110mm Hg at rest
* Symptomatic arterial hypotension
* Known renal artery stenosis
* Serum creatinine > 1.8 mval/l
* Relevant hepatic or pulmonary disorders
* Hyperthyroidism manifested clinically and in laboratory
* Known drug intolerance for AT II inhibitors
* Females who are pregnant or breast feeding
* Females of childbearing potential who are not using a scientifically accepted method of contraception
* Participation in a clinical trial within the last 30 days
* Drug addiction or chronic alcohol abuse
* Legal incapacity, or other circumstances which would prevent the patient from understanding the aim, nature or extent of the clinical study
* Evidence of an uncooperative attitude

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2005-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Percentage of days with documented episodes of paroxysmal atrial fibrillation (number of days with paroxysmal atrial fibrillation/number of days with at least one readable Tele-ECG recording) | 12 months follow-up

SECONDARY OUTCOMES:
Time to first occurrence of a documented relapse of atrial fibrillation | 12 months follow up
Time to first occurrence of a symptomatic documented episode of AF | 12 months follow up
Time to persistent atrial fibrillation | 12 months follow up
Time to prescription of the recovery-medication | 12 months follow up
Number of hospitalizations for cardiovascular reasons (-> Endpoint review) | 12 months follow up
Number of intermediate medical visits for cardiovascular reasons (-> Endpoint review) without hospitalization | 12 months follow up
Number of cerebrovascular events | 12 months follow up
Quality of life | 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meinertz, MD, Principal Investigator — University Hospital Hamburg; Andreas Goette, MD, Principal Investigator — University Hospital Magdeburg

REFERENCES:
- [Derived] von Eisenhart Rothe AF, Goette A, Kirchhof P, Breithardt G, Limbourg T, Calvert M, Baumert J, Ladwig KH. Depression in paroxysmal and persistent atrial fibrillation patients: a cross-sectional comparison of patients enroled in two large clinical trials. Europace. 2014 Jun;16(6):812-9. doi: 10.1093/europace/eut361. Epub 2013 Dec 18. PMID 24351885
- [Derived] von Eisenhart Rothe A, Bielitzer M, Meinertz T, Limbourg T, Ladwig KH, Goette A. Predictors of discordance between physicians' and patients' appraisals of health-related quality of life in atrial fibrillation patients: findings from the Angiotensin II Antagonist in Paroxysmal Atrial Fibrillation Trial. Am Heart J. 2013 Sep;166(3):589-96. doi: 10.1016/j.ahj.2013.05.020. Epub 2013 Jul 10. PMID 24016511
- [Derived] Goette A, Schon N, Kirchhof P, Breithardt G, Fetsch T, Hausler KG, Klein HU, Steinbeck G, Wegscheider K, Meinertz T. Angiotensin II-antagonist in paroxysmal atrial fibrillation (ANTIPAF) trial. Circ Arrhythm Electrophysiol. 2012 Feb;5(1):43-51. doi: 10.1161/CIRCEP.111.965178. Epub 2011 Dec 7. PMID 22157519
- See also: Homepage of the German AF Network — http://www.kompetenznetz-vorhofflimmern.de